CLINICAL TRIAL: NCT00371592
Title: A Phase II, Randomized, Double-blind, Placebo-controlled Trial of Acyclovir for the Suppression of Human Immunodeficiency Virus Type 1 (HIV-1) Viral Load and Mucosal Shedding in HIV-1, Herpes Simplex Virus, Type 2 (HSV-2) Co-Infected Women
Brief Title: Effectiveness of Acyclovir in Suppressing HIV Viral Load in Women Coinfected With HIV and Herpes Simplex Virus Type 2 (HSV-2)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Comprehensive International Program of Research on AIDS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIPRA PE 003; CIPRA Peru Project 1; 10413 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2006-09-01; First posted 2006-09-04 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: HIV Infections; Herpesvirus 2, Human
Keywords: Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Acyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive acyclovir for 24 weeks
  Interventions: Drug: Acyclovir
- 2 (Placebo Comparator): Participants will receive acyclovir placebo for 24 weeks
  Interventions: Drug: Acyclovir placebo

INTERVENTIONS:
Drug: Acyclovir — 800 mg tablet taken orally twice daily
  Other Names: Zovirax
  Arms: 1
Drug: Acyclovir placebo — 800 mg placebo tablet taken orally twice daily
  Other Names: Zovirax placebo
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether acyclovir is effective in suppressing HIV viral load in women infected with both HIV-1 and herpes simplex virus type 2 (HSV-2) who are starting HIV treatment for the first time.

DETAILED DESCRIPTION:
Women coinfected with HIV and HSV-2 experience more genital herpes outbreaks than women infected only with HSV-2. Frequent or recurrent herpes outbreaks in women infected with HIV can lead to an increase in both HIV plasma viral load and cervical shedding of HIV. Some preliminary clinical studies have shown that acyclovir treatment for the management of HSV-2 infection can help lower HIV viral load in patients coinfected with both HIV and HSV-2. Supplementing highly active antiretroviral therapy (HAART) with HSV-2 treatment in patients coinfected with both HIV and HSV-2 may help strengthen the effects of HAART by more effectively lowering plasma and genital HIV viral load. This study will determine whether HSV-2 treatment with acyclovir is effective in controlling HIV plasma viral load and cervical shedding of HIV in women starting on HAART as per Peruvian guidelines.

This study will last 24 weeks. Participants will be randomly assigned into one of two groups. Group 1 participants will receive twice-daily 800 mg of acyclovir for 24 weeks. Group 2 participants will receive twice-daily placebo for 24 weeks. Both groups will receive HAART from the Peruvian Ministry of Health. There will be 15 visits during this study. Medical history; a physical exam; blood collection; family planning counseling; and cervical, vaginal, and vulvar swab collection will begin prior to study entry and will occur at all study visits.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected
* HSV-2 infected
* Initiating HAART per Peruvian guidelines for the first time at study entry
* CD4 count less than 200 cells/mm3 OR CD4 count less than 350 cells/mm3 AND viral load greater than 55,000 copies/ml within 30 days prior to study entry
* Does not intend to move outside of greater metropolitan Lima, Peru area for the duration of the study
* Willing to follow all study requirements
* Willing to provide written informed consent

Exclusion Criteria:

* Prior HAART
* History of adverse reaction to acyclovir, famciclovir, or valacyclovir
* Unwilling to take acyclovir, famciclovir, or valacyclovir
* History of seizures
* Renal insufficiency, defined as serum creatinine greater than 2 mg/dl or a creatinine clearance less than 50 ml/min
* Treatment for a serious medical condition 14 days prior to study entry. Patients with chronic, acute, or recurrent opportunistic infections (OIs) who have completed therapy and are clinically stable on therapy for at least 14 days prior to study entry are not excluded.
* Clinically unstable and untreated OIs or tumors within 14 days prior to study entry. More information on this criterion can be found in the protocol.
* Clinically unstable and untreated bacterial sexually transmitted diseases (STDs) within 14 days prior to study entry. More information on this criterion can be found in the protocol.
* Radiation therapy or systemic chemotherapy within 45 days prior to study entry. Participants who underwent systemic chemotherapy for the treatment of Kaposi's sarcoma (KS) if it was completed prior to study entry are not excluded.
* Any immunomodulator, HIV vaccine, or other investigational therapy within 30 days prior to study entry. Patients who received a tapering course of corticosteroids as acute therapy for Pneumocystis carinii pneumonia (PCP) or are receiving inhaled or nasal fluticasone are not excluded.
* Current drug or alcohol use that, in the investigator's opinion, may interfere with the study
* Vomiting or inability to swallow medications
* Involuntarily incarcerated in a correctional facility, prison, or jail or being detained for the treatment of either a psychiatric or infectious disease
* Grade 2 or 3 high-grade cervical dysplasia and cervical neoplasia within 6 months prior to study entry
* Any other condition that, in the investigator's opinion, may interfere with the study
* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Undetectable HIV plasma RNA viral load (less than 50 copies/ml) | At Week 6

SECONDARY OUTCOMES:
Undetectable HIV plasma RNA viral load (less than 50 copies/ml) | At Week 24
Time to undetectable HIV plasma RNA viral load (less than 50 copies/ml), adjusted for baseline viral load | Throughout study
Intermittent episodes of detectable HIV plasma RNA viral load (greater than 200 copies/ml) | At Weeks 2 and 24
Positive HIV PCR test on vaginal mucosal samples | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Lucchetti, MD, Study Chair — Asociación Civil Impacta Salud y Educación, Lima, Peru; Connie Celum, MD, MPH, Study Chair — University of Washington
Locations (1):
- IMPACTA - San Miguel CIPRA Project 1 CRS, San Miguel, Lima region, Peru

REFERENCES:
- [Background] Posavad CM, Wald A, Kuntz S, Huang ML, Selke S, Krantz E, Corey L. Frequent reactivation of herpes simplex virus among HIV-1-infected patients treated with highly active antiretroviral therapy. J Infect Dis. 2004 Aug 15;190(4):693-6. doi: 10.1086/422755. Epub 2004 Jul 13. PMID 15272395
- [Background] Wright PW, Hoesley CJ, Squires KE, Croom-Rivers A, Weiss HL, Gnann JW Jr. A prospective study of genital herpes simplex virus type 2 infection in human immunodeficiency virus type 1 (HIV-1)-seropositive women: correlations with CD4 cell count and plasma HIV-1 RNA level. Clin Infect Dis. 2003 Jan 15;36(2):207-11. doi: 10.1086/345440. Epub 2003 Jan 6. PMID 12522754
- [Background] Schacker T, Zeh J, Hu H, Shaughnessy M, Corey L. Changes in plasma human immunodeficiency virus type 1 RNA associated with herpes simplex virus reactivation and suppression. J Infect Dis. 2002 Dec 15;186(12):1718-25. doi: 10.1086/345771. Epub 2002 Nov 22. PMID 12447756